CLINICAL TRIAL: NCT04961892
Title: Difference of Plantar Pressure Distribution Between Surgical Treatment and Conservative Treatment for Chronic Ankle Instability
Brief Title: Difference of Plantar Pressure Distribution Between Surgical Treatment and Conservative Treatment for CAI
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019164
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Chronic Ankle Instability
MeSH Terms: interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgical treatment: Patients with CAI undergoing surgical treatment
  Interventions: Procedure: surgical treatment
- conservative treatment: Patients with CAI undergoing conservative treatment
  Interventions: Procedure: conservative treatment

INTERVENTIONS:
Procedure: surgical treatment — Anatomical contraction and termination reconstruction of the lateral ligament
  Groups: surgical treatment
Procedure: conservative treatment — Rehabilitation intervention training
  Groups: conservative treatment

SUMMARY:
The objective of this study was to compare the difference of plantar pressure distribution between surgical treatment and conservative treatment for CAI.

DETAILED DESCRIPTION:
The data of 20 patients who underwent surgery after reconstruction of the lateral collateral ligament of the ankle joint and 20 patients who underwent balance rehabilitation training were analyzed to compare the clinical effects of surgical treatment and conservative treatment for chronic ankle instability, in order to better guide the selection of the optimal intervention program for patients with chronic ankle joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CAI
* The contralateral ankle joint is healthy

Exclusion Criteria:

* Accompanied by other musculoskeletal injuries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From April 1, 2019, information of 20 patients diagnosed with CAI that underwent surgical treatment in our institute and 20 patients that underwent conservative treatment was collected and evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
FAAM | pre-surgery, one year after sugery
  Foot and Ankle Ability Measure Activity

SECONDARY OUTCOMES:
IDFAI | pre-surgery, one year after sugery
  Identification of Functional Ankle Instability questionnaire
Ligament injury by MRI | pre-surgery, one year after sugery
  To evaluate the condition of lateral collateral ligament using magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Yuelin Hu, bachelor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No